CLINICAL TRIAL: NCT01328223
Title: Phase II Study of Combined Sorafenib With Radiotherapy in Patients With Advanced Hepatocellular Carcinoma
Brief Title: Study of Combined Sorafenib With Radiotherapy in Patients With Advanced Hepatocellular Carcinoma
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: China Medical University Hospital (Other)
Responsible Party: Shang-Wen Chen, Department of Radiation Oncology
Other Study IDs: Radiotherapy-Sorafenib
Record Dates: First submitted 2011-03-20; First posted 2011-04-04 (Estimated); Last update posted 2011-04-04 (Estimated); Status verified 2011-03

CONDITIONS: Hepatocellular Carcinoma
Keywords: Hepatocellular carcinoma; radiotherapy; sorafenib
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Sorafenib; Radiotherapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- radiotherapy efficacy: 1. Concurrent stage with RT: sorafenib 400mg twice daily
  2. Maintenance stage after RT: sorafenib 400mg twice daily Treatment can be continued until the occurrence of clinical or radiologic progression, the occurrence of either unacceptable adverse events, death, or any criteria met for removal from the protocol treatment. Basically, minimum maintenance duration of 6 months is recommended, not mandatory.
  Interventions: Radiation: sorafenib and radiotherapy for hepatocellular carcinoma

INTERVENTIONS:
Radiation: sorafenib and radiotherapy for hepatocellular carcinoma — Concurrent and maintenance sorafenib 400mg twice daily
  Other Names: Combined radiotherapy and sorafenib.

SUMMARY:
Hepatocellular carcinoma (HCC) is a common cause of cancer mortality in Asia. Most patients present with intermediate or advanced disease. Percutaneous ethanol injection, radiofrequency ablation, and transcatheter arterial chemoembolization (TACE) are not considered as a curative treatment and have achieved very limited success in eradicating large HCC. With the development of new radiotherapy (RT) technique, RT can be more safely given to patients with larger tumor burden. Thus, TACE combined with RT has been suggested for treating large HCC. Based on the results of these studies, RT could achieve a tumor response rate of 50 % to 70 %. However, it has not been definitively shown to prolong the overall or disease-free survival due to lack of a phase III clinical trial. In contrast, a retrospective clinical investigation with molecular study suggests that sublethal dose of RT promoted HCC growth outside RT field.

Two phase III trials were shown to be efficacious and well-tolerated in patients with advanced HCC. Median overall survival was significantly 2 to 3 months longer in the sorafenib group than that in the placebo. It is interesting to recognize the combined therapeutic effect of RT with sorafenib. Based on several preclinical experiments, tumor angiogenesis inhibitors seem to be synergistic with irradiation when using before RT, concurrently with RT, or after RT. Thus, the investigators design a single-arm phase II clinical trial to investigate the efficacy of combined RT with sorafenib.

The eligibility criteria are patients with unresectable HCC; good performance status; no prior radiotherapy for the liver; clinical measurable tumor; good liver function and good compliance. After entering this study, the testee will receive RT to hepatic tumor with concurrently sorafenib with a dose of 400 mg twice daily. Hepatic RT will be performed with a daily fraction size of 2.0 to 2.5 Gy to a total dose of 46 Gy to 60 Gy. After RT, maintenance sorafenib with a dose of 400 mg twice daily will be ongoing. Sorafenib will be continued until the occurrence of clinical or radiologic progression, or the occurrence of either unacceptable adverse events or death. Minimum maintenance duration of 6 months is recommended, but not mandatory.

DETAILED DESCRIPTION:
The primary end points are response rate and toxicities profile. The secondary endpoints are time to disease-free survival, overall survival, and quality of life assessment.

ELIGIBILITY:
Inclusion Criteria:

* Patients with unresectable hepatoma with transarterial embolization (TAE) failure or who are not suitable for TACE. A maximal tumor diameter > 3.0 cm.
* Age: 20 ~ 69 years.
* ECOG 0 or 1.
* Life expectancy of at least 12 weeks.
* Child-Pugh A or B (preferentially score ≦ 7).
* Cancer of the Liver Italian Program (CLIP) score ≦ 3.
* Pretreatment liver function test and renal function test:

  * Total bilirubin < 1.5 times the upper limit of normal (ULN)(≦ 3.0 (ULN) in patients treated by biliary drainage for obstructive jaundice)
  * GOP/GPT ≦ 5 X of upper limit of normal range
  * Alkaline phosphatase ≦ 4X of upper limit of normal range
  * Prothrombin time/partial prothrombin time < 1.5 X of ULN
  * Serum Creatinine ≦ 1.0 x ULN
* Pretreatment blood count:

  * Hemoglobulin ≧ 9 g/dl
  * Absolute neutrophil count ≧ 1500/mm3
  * Platelet count ≧ 50,000/mm3
* Subjects with at least one uni-dimensional or bi-dimensional measurable lesion. Lesion must be measured by CT scan or MRI.
* Patients must fully recover from prior therapy that given > 4 weeks before enrollment.
* Signed informed consent must be obtained prior to any study related procedures.

Exclusion Criteria:

1. Child-Pugh C
2. CLIP score ≧ 4
3. Patients with evidence of extrahepatic or metastatic disease
4. Patients with evidence of massive ascites
5. Patients receiving previous irradiation to liver
6. Patients with previous use of Thalidomide less than 6 months from entering of the study
7. History of cardiac disease: congestive heart failure >NYHA class 2; active CAD (MI more than 6 mo prior to study entry is allowed); cardiac arrythmias requiring anti-arrythmic therapy (beta blockers or digoxin are permitted)
8. Active clinically serious infections ( > grade 2 CTC version 2)
9. Patients undergoing renal dialysis
10. Patients with evidence or history of bleeding diathesis
11. Prior treatment with EGFR TKIs or VEGFR TKIs
12. Hypertension uncontrolled by medical therapy
13. Symptomatic metastatic brain or meningeal tumors unless the patient is > 6 months from definitive therapy, has a negative imaging study within 4 weeks of study entry and is clinically stable with respect to the tumor at the time of study entry. Also the patient must not be undergoing acute steroid therapy or taper.
14. Chemotherapy or immunotherapy or other systemic anti-cancer therapy within 4 weeks.

Ages: 20 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Paitents with unresectable hepatoma with transarterial chemoembolization (TACE) failure or who are not suitable for TACE.
Sampling Method: Non-Probability Sample
Enrollment: 45 (Estimated)
Dates: Start 2010-09; Primary Completion 2012-06 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
Response rate | 6 months
  1. The tumor response rate will be evaluated at the 6th month after the ending of radiotherapy.
  2. The response rate includes complete and partial response according to the RECIST (Response Evaluation Criteria in Solid Tumors) criteria.

SECONDARY OUTCOMES:
Disease progression-free survival | 2 years
  Disease progression-free survival:
  Patients with the evidence of clinical or radiographic progressive disease will be defined as disease progression. The average time period for the follow-up will be two years.
Overall survival | 2 years
  Participants will be followed. The average time period will be two years.

CONTACTS AND LOCATIONS:
Overall Officials: Shang-Wen Chen, MD, Principal Investigator — Department of Radiation Oncology, China Medical University Hospital
Locations (3):
- Taiwan (3):
  - Shang-Wen Chen, Taichung, Taiwan
  - Li-Ching Lin, Tainan, Taiwan
  - Jeng-Fong Chiou, Taipei, Taiwan